CLINICAL TRIAL: NCT06814470
Title: A Feasibility Study of Virtual Reality Guided Acupuncture Imagery Treatment for Chronic Low Back Pain
Brief Title: Virtual Reality Guided Acupuncture Imagery Treatment for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lucy Chen, Principal investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018p002553-1
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2024-11

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Intervention Model Description: subject will be randomized to 2 groups
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality - guided acupuncture imagery treatment (VRGAIT) (Experimental)
  Interventions: Other: Virtual reality guided imagery acupuncture treatment (VRGAIT)
- Virtual Reality -guided acupuncture imagery treatment (VRGAIT) Control (Active Comparator)
  Interventions: Other: Virtual reality guided imagery acupuncture treatment control

INTERVENTIONS:
Other: Virtual reality guided imagery acupuncture treatment (VRGAIT) — Subject watching Virtual reality video of acupuncture needle stimulation
  Arms: Virtual Reality - guided acupuncture imagery treatment (VRGAIT)
Other: Virtual reality guided imagery acupuncture treatment control — Subject watching VR video of swab touching
  Arms: Virtual Reality -guided acupuncture imagery treatment (VRGAIT) Control

SUMMARY:
Testing the effect of Virtual Reality - guided imagery acupuncture

DETAILED DESCRIPTION:
The aim of this study is to develop a Virtual Reality guided acupuncture imagery treatment system for the treatment of chronic low back pain. This product will provide a new cost-effective treatment option for chronic low back pain and potentially other chronic pain disorders.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers 18-75 years of age.
* Meet the Classification Criteria of chronic LBP (having low back pain for more than 6 months), as determined by the referring physician.
* At least 4/10 clinical pain on the 11-point LBP intensity scale.
* Must have had a prior evaluation of their low back pain by a health care provider, which may have included radiographic studies. Documentation of this evaluation will be sought from Partners or outside medical records and kept in the subject's research record.
* At least a 10th grade English-reading level; English can be a second language provided that the patients feel they understand all the questions used in the assessment measures.

Exclusion Criteria:

* Specific causes of back pain (e.g. cancer, fractures, infections),
* Complicated back problems (e.g. prior back surgery, medico legal issues),
* Possible contraindications for acupuncture (e.g. coagulation disorders, cardiac pacemakers, pregnancy, seizure disorder), and conditions that might confound longitudinal effects or interpretation of results (e.g. severe fibromyalgia, rheumatoid arthritis).
* Conditions making study participation difficult (eg, paralysis, psychoses, or other severe psychological problems as per the judgment of a study investigator during Session 1)
* The intent to undergo surgery during the time of involvement in the study.
* Unresolved medical legal/disability/workers compensation claims in connection with low back pain.
* Lacking the capacity to consent for oneself
* Do not have access to zoom or other software regularly to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lucy Chen, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The Small Business Act permits NIH SBIR/STTR grantees to withhold data for 4 years after the end of the grant award.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Reality - Guided Acupuncture Imagery Treatment (VRGAIT) | Virtual Reality -Guided Acupuncture Imagery Treatment (VRGAIT) Control
Started | 15 | 16
Completed | 14 | 14
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Individuals with chronic low back pain
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality - Guided Acupuncture Imagery Treatment (VRGAIT) | Virtual Reality -Guided Acupuncture Imagery Treatment (VRGAIT) Control | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: year] | 48 (16) | 50 (17) | 49 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 8 | 10 | 18
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Proportion of subjects who complete all assessments from the total number of subjects who were enrolled in the study
Time Frame: Through study intervention, an average of about four weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality - Guided Acupuncture Imagery Treatment (VRGAIT) | Virtual Reality -Guided Acupuncture Imagery Treatment (VRGAIT) Control
Number analyzed (Participants) | 15 | 16
Participants | 14 | 14

2. Primary Outcome: Satisfaction to the Interventions
Description: Mean of the satisfaction score on a scale from 1 to 5, larger number indicated greater satisfaction. Assessed after each study interventions, an average score is reported.,
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Virtual Reality - Guided Acupuncture Imagery Treatment (VRGAIT) | Virtual Reality -Guided Acupuncture Imagery Treatment (VRGAIT) Control
Number analyzed (Participants) | 14 | 14
scores on a scale | 4.7 (.33) | 3.9 (1.0)

3. Primary Outcome: Number of Adverse Events (Safety of the Intervention)
Description: Symptoms and adverse events reported by the participants
Time Frame: Through study interventions, an average of about four weeks
Measure: Number; unit: number of adverse event
Arm/Group | Virtual Reality - Guided Acupuncture Imagery Treatment (VRGAIT) | Virtual Reality -Guided Acupuncture Imagery Treatment (VRGAIT) Control
Number analyzed (Participants) | 15 | 16
number of adverse event | 0 | 0

4. Secondary Outcome: PROMIS-29
Description: The PROMIS-29 profile measure assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items for each domain. We use pain intensity in this report, low score indicates improvement.
Time Frame: baseline, midpoint (week 2), and post-treatment (week 4), the change of score (baseline minus post-treatment) is reported.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Virtual Reality - Guided Acupuncture Imagery Treatment (VRGAIT) | Virtual Reality -Guided Acupuncture Imagery Treatment (VRGAIT) Control
Number analyzed (Participants) | 14 | 14
scores on a scale | 1 [0.2 to 1.8] | 0.5 [.3 to 1.3]

5. Secondary Outcome: Pain Bothersomeness Scale
Description: This is a self-reported measure of cLBP pain severity that is commonly used to assess clinical chronic pain. Participants rate how bothersome their LBP was during the previous week with a VAS scale (0-10) from "not at all bothersome" (0) to "extremely bothersome" (10).
Time Frame: as for outcome 4
Population: pre minus post intervention score is reported
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Virtual Reality - Guided Acupuncture Imagery Treatment (VRGAIT) | Virtual Reality -Guided Acupuncture Imagery Treatment (VRGAIT) Control
Number analyzed (Participants) | 14 | 14
scores on a scale | 2 [0.8 to 3.2] | 0.71 [0.5 to 1.9]

6. Secondary Outcome: MGH Acupuncture Sensation Scale (MASS)
Description: MASS is a scale developed to measure sensations evoked by acupuncture treatment (total range 0-120). The MASS will be applied after each treatment. We reported total score in this report (average of sum of each session). larger numbers indicate stronger sensations.
Time Frame: up to 4 weeks.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Virtual Reality - Guided Acupuncture Imagery Treatment (VRGAIT) | Virtual Reality -Guided Acupuncture Imagery Treatment (VRGAIT) Control
Number analyzed (Participants) | 14 | 14
unit on a scale | 9.0 (10.0) | 4.5 (5.3)

7. Secondary Outcome: Vividness Scale
Description: Vividness Scale is a 0-10 vividness scale to measure imagery vividness during the intervention. The scale ranges from Not Vivid/Unclear (0) to Vivid/Clear (10).
Time Frame: After each study interventions, the average score is reported.
Measure: Mean (Standard Deviation); unit: the unit on the scale
Arm/Group | Virtual Reality - Guided Acupuncture Imagery Treatment (VRGAIT) | Virtual Reality -Guided Acupuncture Imagery Treatment (VRGAIT) Control
Number analyzed (Participants) | 14 | 14
the unit on the scale | 8.6 (1.7) | 7.9 (2.0)

ADVERSE EVENTS:
Time Frame: 1 months
Arm/Group | Virtual Reality - Guided Acupuncture Imagery Treatment (VRGAIT) | Virtual Reality -Guided Acupuncture Imagery Treatment (VRGAIT) Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT06814470/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT06814470/SAP_001.pdf